CLINICAL TRIAL: NCT01577537
Title: A Phase 3, Double-blind, Multicentre, Randomised, Placebo-controlled Study to Assess the Efficacy and Safety of SPL7013 Gel (VivaGel) for the Treatment of Bacterial Vaginosis
Brief Title: A Phase 3 Study of SPL7013 Gel (VivaGel) for the Treatment of Bacterial Vaginosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Starpharma Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPL7013-016
Record Dates: First submitted 2012-04-12; First posted 2012-04-16 (Estimated); Results first posted 2019-07-09 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Bacterial Vaginosis
Keywords: SPL7013; VivaGel; bacterial vaginosis; BV
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — astodrimer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VivaGel (Experimental)
  Interventions: Drug: 1% SPL7013 Gel
- HEC Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 1% SPL7013 Gel — Vaginal gel, daily for 7 days
  Other Names: VivaGel
  Arms: VivaGel
Drug: Placebo — Vaginal gel, daily for 7 days
  Arms: HEC Placebo

SUMMARY:
The primary objective of the study is to assess the efficacy of 1% SPL7013 Gel compared to placebo gel for the treatment of bacterial vaginosis (BV).

After screening eligible participants will be randomized to receive either 1% SPL7013 Gel or hydroxyethyl cellulose (HEC) placebo gel at a dose of 5g administered vaginally at bedtime for 7 consecutive days. Participants will be assessed for BV (both by Amsel criteria and Nugent score) at screening/Baseline, after last application (End of Treatment, EOT, Day 9-12) and at the final study visit approximately 2-3 weeks after last dose (Test of Cure, TOC, Day 21-30).

ELIGIBILITY:
Key eligibility criteria:

* Post-menarchal females, aged 12 years or more
* Diagnosis of BV by Amsel criteria (ie all four of the following signs/symptoms: presence of white to grey homogeneous discharge; positive whiff test indicating an amine (fishy) odor with addition of potassium hydroxide; vaginal pH greater than 4.5; and presence at least 20% clue cells of total epithelial cells
* Nugent score of at least 4
* Otherwise healthy, as determined by medical history, physical examination
* normal Pap smear at or documented within 24 months of screening

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2012-04-17 (Actual); Primary Completion 2012-10-05 (Actual); Study Completion 2012-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Paull, PhD, Study Chair — Starpharma Pty Ltd

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VivaGel | HEC Placebo
Started | 128 | 123
Completed | 120 | 116
Not Completed | 8 | 7

BASELINE CHARACTERISTICS:
Population: modified intent-to-treat (mITT) population, which included all participants in the Safety population who had a Nugent score of 4-10 at Baseline, but excluded those with a Nugent score of 0-3.
Groups:
- Total: Total of all reporting groups
Arm/Group | VivaGel | HEC Placebo | Total
Number analyzed (Participants) | 120 | 117 | 237
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (9.9) | 36.2 (12.3) | 35.6 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 117 | 237
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 83 | 81 | 164
  Belgium | 10 | 10 | 20
  Germany | 27 | 26 | 53

OUTCOME MEASURES:

1. Primary Outcome: Number of Women With Clinical Cure at the End of Treatment Visit (EOT)
Description: Clinical Cure is defined as the resolution of clinical findings (ie Amsel criteria) from the Baseline visit (Day 1)
Time Frame: Day 9-12
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | VivaGel | HEC Placebo
Number analyzed (Participants) | 120 | 117
Participants | 68 | 25
Statistical Analysis 1: Comparison: VivaGel vs HEC Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel

2. Secondary Outcome: Number of Women With Nugent Cure at the EOT Visit
Description: Nugent Cure is defined as a Nugent score of 0-3 (normal)
Time Frame: Day 9-12
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | VivaGel | HEC Placebo
Number analyzed (Participants) | 120 | 117
Participants | 16 | 6

3. Secondary Outcome: Number of Women With Clinical Cure at the Test of Cure Visit (TOC)
Description: Clinical Cure is defined as the resolution of clinical findings (ie Amsel criteria) from the Baseline visit (Day 1)
Time Frame: Day 21-30
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | VivaGel | HEC Placebo
Number analyzed (Participants) | 120 | 117
Participants | 34 | 33

4. Secondary Outcome: Number of Women With Nugent Cure at the TOC Visit
Description: Nugent Cure is defined as a Nugent score of 0-3 (normal)
Time Frame: Day 21-30
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | VivaGel | HEC Placebo
Number analyzed (Participants) | 120 | 117
Participants | 16 | 13

5. Secondary Outcome: Adverse Events Potentially Related to Treatment
Description: Number of participants experiencing adverse events considered potentially related to study treatment.
Time Frame: Screening/baseline through TOC visit, Day 1-30
Population: Safety population. Two participants of those randomized to the 1% SPL7013 Gel group withdrew consent, did not use study medication, and therefore were not included in the Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | VivaGel | HEC Placebo
Number analyzed (Participants) | 126 | 123
Participants | 17 | 9

ADVERSE EVENTS:
Description: Analysis of all participants who received (were dispensed) the study medication, excluding any participants who returned all the study medication unused (Safety population). This population is broader than the modified intent-to-treat population, which included all participants in the Safety population who had a Nugent score of 4-10 at Baseline, but excluded those with a Nugent score of 0-3.
Arm/Group | VivaGel | HEC Placebo
Serious Adverse Events (participants affected / at risk) | 0/126 | 0/123
Other Adverse Events (participants affected / at risk) | 0/126 | 0/123

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For multicenter studies, PIs can publish only after data from all sites are published collectively.